CLINICAL TRIAL: NCT03784300
Title: A Phase I, Single Center, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose, Pharmacokinetic and Safety Study of PTl-125 in Healthy Volunteers
Brief Title: A Safety Study of PTI-125 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pain Therapeutics (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: Cassava Sciences, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PTI-125-01; 1R44AG056166 (NIH)
Record Dates: First submitted 2018-12-18; First posted 2018-12-21 (Actual); Results first posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Alzheimer Disease, Early Onset; Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Simufilam

STUDY DESIGN:
Intervention Model Description: Single center, randomized, double-blind, placebo controlled, SAD study of three escalating doses of PTI-125. A total of 24 healthy subjects enrolled in one of three dose cohorts. Each cohort will contain 8 subjects; six receive PTI-125 and two receive placebo. Three SAD does of PTI-125 oral solution (50, 100 or 200 mg) or placebo solution will be administered.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 50 mg PTI-125 (Active Comparator): Six (6) subjects will receive a single orally administered dose of 50 mg PTI-125 in this cohort.
  Interventions: Drug: 50 mg PTI-125
- 50 mg PTI-125 Placebo (Placebo Comparator): Two (2) subjects will receive a single orally administered dose of 50 mg Placebo PTI-125 in this cohort.
  Interventions: Drug: 50 mg PTI-125
- 100 mg PTI-125 (Active Comparator): Six (6) subjects will receive a single orally administered dose of 100 mg PTI-125 in this cohort.
  Interventions: Drug: 100 mg PTI-125
- 100 mg PTI-125 Placebo (Placebo Comparator): Two (2) subjects will receive a single orally administered dose of 100 mg Placebo PTI-125 in this cohort.
  Interventions: Drug: 100 mg PTI-125
- 200 mg PTI-125 (Active Comparator): Six (6) subjects will receive a single orally administered dose of 200 mg PTI-125 in this cohort.
  Interventions: Drug: 200 mg PTI-125
- 200 mg PTI-125 Placebo (Placebo Comparator): Two (2) subjects will receive a single orally administered dose of 200 mg Placebo PTI-125 in this cohort.
  Interventions: Drug: 200 mg PTI-125

INTERVENTIONS:
Drug: 50 mg PTI-125 — PTI-125 50 mg Oral Solution
  Arms: 50 mg PTI-125; 50 mg PTI-125 Placebo
Drug: 100 mg PTI-125 — PTI-125 100 mg Oral Solution
  Arms: 100 mg PTI-125; 100 mg PTI-125 Placebo
Drug: 200 mg PTI-125 — PTI-125 200 mg Oral Solution
  Arms: 200 mg PTI-125; 200 mg PTI-125 Placebo

SUMMARY:
A Phase I, Single Center, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose, Pharmacokinetic and Safety Study of PTl-125 in Healthy Volunteers

DETAILED DESCRIPTION:
This was a Phase I, single center, randomized, double-blind, placebo-controlled, single ascending dose (SAD) study in healthy volunteers, 18 to 45 years of age. A total of twenty-four (24) subjects were enrolled into the study in one of three dose cohorts. Each cohort contained eight subjects; six subjects received PTI-125 and two received placebo. Three doses of PTI-125 oral solution (50, 100, and 200 mg) or placebo solution were administered to respective cohorts.

The study included a screening period (Day -28 to Day -1), an inpatient treatment period (Day 0 through Day 4), and a follow-up visit (Day 7). Subjects reported to the clinic on the day before dosing and were randomized to receive either a single dose of orally administered PTI-125 or placebo. Each dose was administered following an overnight fast of at least 10 hours.

For each dose level, dosing was staggered such that two subjects (one active and one placebo) were dosed prior to the rest of the group. After a minimum of 24 hours and review of all 24-hour safety assessments (electrocardiogram [ECG], a brief physical examination, vital signs, and laboratory assessments) an independent Data Safety Monitoring Board/Data Monitoring Committee (DSMB/DMC) determined whether the remaining 6 subjects were to be dosed.

Pharmacokinetic blood samples were obtained prior to dosing and at specified intervals during the study (0-72 hours post-dose). Blood draws for laboratory testing were performed prior to dosing and at 24 hours post dose. After safety assessments of ECG, vital signs, and a brief physical exam at 72 hours, subjects were discharged from the clinic and returned 7 days post-dose for a final safety assessment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 18 and 45 years of age, inclusive.
* The subject has a body mass index (BMI) within 18-30 kg/m2 (inclusive).
* The subject is in good health as determined by medical history and physical examination and clinical laboratory parameters.
* The subject is willing and able to speak, read, and understand English and provide written informed consent.
* The subject is a non-smoker for at least 12 months. If a former smoker, the reason for stopping must be evaluated.
* Females who are physically incapable of childbearing defined as postmenopausal, or surgically sterile (hysterectomy, bilateral tubal ligation, bilateral oophorectomy or an Essure procedure). Appropriate documentation (ex; medical record) of the surgical sterilization procedure to be obtained and held within the subject's study file.
* The subject must agree to comply with the drawing of blood samples for the PK assessments.
* The subject is willing and able to comply with all testing and requirements defined in the protocol.
* The subject is willing and able to remain at the study site unit for the duration of the confinement period and return for the outpatient visit.

Exclusion Criteria:

* The subject has any relevant deviations from normal in physical examination, electrocardiogram (ECG), or clinical laboratory tests, as evaluated by the investigator.
* The subject has had a clinically significant illness within 30 days of Check-in.
* The subject has a history of significant neurological, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, or metabolic disease.
* The subject has used any prescription medication within 14 days of dosing or overthe- counter (OTC) medication within 48 h of dosing or intends to use any prescription medication or OTC medication during the study that may interfere with the evaluation of study medication.
* The subject has used alcohol, caffeine or xanthine-containing products 48 h before dosing or intends to use any of these products during the study.
* The subject has used grapefruit, grapefruit juice, or grapefruit-containing products days before dosing or intends to use any of these products during the study.
* The subject has a history of substance abuse or a positive ethanol breath test, urine cotinine, or urine drug screen at screening or at check-in. The subject has a positive serum hepatitis B surface antigen or positive HCV antibody test at the Screening Visit.
* The subject has a positive HIV test at the Screening Visit.
* Female subject is pregnant or breastfeeding.
* The subject has received an investigational drug within 30 days of Check-in.
* The subject has donated or lost a significant volume of blood (>450 mL) within 4 weeks prior to the study.
* The subject is unwilling to reside in the study unit for the duration of the study or to cooperate fully with the investigator or site personnel.
* The subject has an AST/ALT or total bilirubin greater than the ULN. One repeat test will be allowed.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2017-10-09 (Actual); Study Completion 2018-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George J Atiee, MD, Principal Investigator — Worldwide Clinical Trials
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 50 mg PTI-125 | 50 mg PTI-125 Placebo | 100 mg PTI-125 | 100 mg PTI-125 Placebo | 200 mg PTI-125 | 200 mg PTI-125 Placebo
Started | 6 | 2 | 6 | 2 | 6 | 2
Completed | 6 | 2 | 6 | 2 | 6 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 50 mg PTI-125 | 50 mg PTI-125 Placebo | 100 mg PTI-125 | 100 mg PTI-125 Placebo | 200 mg PTI-125 | 200 mg PTI-125 Placebo | Total
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 2 | 6 | 2 | 6 | 2 | 24
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: Years] | 38.2 [18 to 45] | 31.8 [18 to 45] | 35.3 [18 to 45] | 31.8 [18 to 45] | 35.8 [18 to 45] | 31.8 [18 to 45] | 35.3 [18 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 0 | 1 | 0 | 4
  Male | 4 | 2 | 5 | 2 | 5 | 2 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 4 | 2 | 2 | 1 | 13
  White | 3 | 1 | 2 | 0 | 4 | 1 | 11
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 2 | 6 | 2 | 6 | 2 | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The peak drug concentration will be obtained directly from the data without interpolation.
Time Frame: Blood samples will be drawn on Day 1 after dosing at 20, 40, and 60 minutes and at 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours.
Population: Separate dose cohorts of 6 active and 2 placebo received 50, 100, or 200 mg. A sentinel dose group of 1 active and 1 placebo preceded each full dose cohort.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 50 mg PTI-125 | 50 mg PTI-125 Placebo | 100 mg PTI-125 | 100 mg PTI-125 Placebo | 200 mg PTI-125 | 200 mg PTI-125 Placebo
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2
ng/mL | 315 (96.6) | NA (NA) — Pk values N/A for placebo subjects | 550 (146) | NA (NA) — Pk values N/A for placebo subjects | 1240 (276) | NA (NA) — Pk values N/A for placebo subjects

2. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) (Tmax)
Description: The time to peak drug concentration will be obtained directly from the data without interpolation
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 50 mg PTI-125 | 50 mg PTI-125 Placebo | 100 mg PTI-125 | 100 mg PTI-125 Placebo | 200 mg PTI-125 | 200 mg PTI-125 Placebo
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2
hours | 1.56 (0.69) | NA (NA) — Pk values N/A for placebo subjects | 1.08 (0.48) | NA (NA) — Pk values N/A for placebo subjects | 1.28 (0.57) | NA (NA) — Pk values N/A for placebo subjects

3. Primary Outcome: Time to Last Quantifiable Plasma Concentration (Tlast)
Description: The time to the last quantifiable drug concentration will be obtained directly from the data without interpolation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 50 mg PTI-125 | 50 mg PTI-125 Placebo | 100 mg PTI-125 | 100 mg PTI-125 Placebo | 200 mg PTI-125 | 200 mg PTI-125 Placebo
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2
hours | 44.0 (16.4) | NA (NA) — Pk values N/A for placebo subjects | 46.0 (4.6) | NA (NA) — Pk values N/A for placebo subjects | 50.00 (11.8) | NA (NA) — Pk values N/A for placebo subjects

4. Primary Outcome: Last Quantifiable Plasma Concentration (Clast)
Description: The concentration of the last quantifiable drug will be obtained directly from the data without interpolation concentration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 50 mg PTI-125 | 50 mg PTI-125 Placebo | 100 mg PTI-125 | 100 mg PTI-125 Placebo | 200 mg PTI-125 | 200 mg PTI-125 Placebo
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2
ng/mL | 1.04 (0.495) | NA (NA) — Pk values N/A for placebo subjects | 0.795 (0.294) | NA (NA) — Pk values N/A for placebo subjects | 0.806 (0.292) | NA (NA) — Pk values N/A for placebo subjects

5. Primary Outcome: Elimination Rate Constant (λz)
Description: The elimination rate constant (λz) will be calculated.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | 50 mg PTI-125 | 50 mg PTI-125 Placebo | 100 mg PTI-125 | 100 mg PTI-125 Placebo | 200 mg PTI-125 | 200 mg PTI-125 Placebo
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2
1/hour | 0.141 (0.0539) | NA (NA) — Pk values N/A for placebo subjects | 0.157 (0.0155) | NA (NA) — Pk values N/A for placebo subjects | 0.144 (0.0516) | NA (NA) — Pk values N/A for placebo subjects

6. Primary Outcome: Termination Elimination Half-Life (T1/2)
Description: The terminal elimination half-life (T1/2) will be calculated.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 50 mg PTI-125 | 50 mg PTI-125 Placebo | 100 mg PTI-125 | 100 mg PTI-125 Placebo | 200 mg PTI-125 | 200 mg PTI-125 Placebo
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2
hours | 6.05 (3.87) | NA (NA) — Pk values N/A for placebo subjects | 4.45 (0.39) | NA (NA) — Pk values N/A for placebo subjects | 5.93 (3.87) | NA (NA) — Pk values N/A for placebo subjects

7. Primary Outcome: Area Under the Curve (AUC)
Description: The AUC from time zero to the time of the last quantifiable concentration (AUClast) will be calculated.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 50 mg PTI-125 | 50 mg PTI-125 Placebo | 100 mg PTI-125 | 100 mg PTI-125 Placebo | 200 mg PTI-125 | 200 mg PTI-125 Placebo
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2
h*ng/mL | 2040 (893) | NA (NA) — Pk values N/A for placebo subjects | 3130 (1150) | NA (NA) — Pk values N/A for placebo subjects | 8130 (1530) | NA (NA) — Pk values N/A for placebo subjects

8. Primary Outcome: Area Under the Curve to Infinity (AUCinf)
Description: The AUC from time zero extrapolated to infinity (AUCinf) will be calculate.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 50 mg PTI-125 | 50 mg PTI-125 Placebo | 100 mg PTI-125 | 100 mg PTI-125 Placebo | 200 mg PTI-125 | 200 mg PTI-125 Placebo
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2
h*ng/mL | 2180 (897) | NA (NA) — Pk values N/A for placebo subjects | 3260 (1150) | NA (NA) — Pk values N/A for placebo subjects | 8250 (1530) | NA (NA) — Pk values N/A for placebo subjects

9. Primary Outcome: Percent Extrapolated of Area Under the Curve to Infinity (AUCextrap[%]).
Description: The percentage of AUCinf based on extrapolation (AUCextrap[%]).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent extrapolated
Arm/Group | 50 mg PTI-125 | 50 mg PTI-125 Placebo | 100 mg PTI-125 | 100 mg PTI-125 Placebo | 200 mg PTI-125 | 200 mg PTI-125 Placebo
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2
percent extrapolated | 0.410 (0.187) | NA (NA) — Pk values N/A for placebo subjects | 0.151 (0.0366) | NA (NA) — Pk values N/A for placebo subjects | 0.144 (0.0156) | NA (NA) — Pk values N/A for placebo subjects

10. Primary Outcome: Oral Clearance (Cl/F)
Description: The apparent oral clearance will be calculated.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: (L/h)
Arm/Group | 50 mg PTI-125 | 50 mg PTI-125 Placebo | 100 mg PTI-125 | 100 mg PTI-125 Placebo | 200 mg PTI-125 | 200 mg PTI-125 Placebo
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2
(L/h) | 25.7 (8.42) | NA (NA) — Pk value not available as these are placebo patients | 33.0 (8.16) | NA (NA) — Pk value not available as these are placebo patients | 24.9 (4.53) | NA (NA) — Pk value not available as these are placebo patients

11. Primary Outcome: Volume of Distribution (Vz/F)
Description: Vz/F, apparent volume of distribution will be calculated.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: (L)
Arm/Group | 50 mg PTI-125 | 50 mg PTI-125 Placebo | 100 mg PTI-125 | 100 mg PTI-125 Placebo | 200 mg PTI-125 | 200 mg PTI-125 Placebo
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2
(L) | 199 (64.9) | NA (NA) — Pk value not available as these are placebo patients | 215 (64.8) | NA (NA) — Pk value not available as these are placebo patients | 214 (154) | NA (NA) — Pk value not available as these are placebo patients

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | 50 mg PTI-125 | 50 mg PTI-125 Placebo | 100 mg PTI-125 | 100 mg PTI-125 Placebo | 200 mg PTI-125 | 200 mg PTI-125 Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2
Other Adverse Events (participants affected / at risk) | 0/6 | 0/2 | 1/6 | 0/2 | 1/6 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50 mg PTI-125 (N=6) | 50 mg PTI-125 Placebo (N=2) | 100 mg PTI-125 (N=6) | 100 mg PTI-125 Placebo (N=2) | 200 mg PTI-125 (N=6) | 200 mg PTI-125 Placebo (N=2)
lightheadedness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — lightheadedness upon standing was resported for a subject in the 100 mg group at 1 h post-dose
transient musculoskeletal wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — One subject in the 200 mg group reported transient musculoskeletal wall pain
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — The same subject in the 200 mg group who reported transient musculoskeletal wall pain, also reported acne

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT03784300/Prot_SAP_ICF_000.pdf